CLINICAL TRIAL: NCT01580098
Title: Regions of Europe Working Together for Health (Renewing Health)
Brief Title: Medium-term Health Coaching and Life-long Monitoring in Diabetes Mellitus
Acronym: RenewingHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landeskrankenanstalten-Betriebsgesellschaft (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D250487
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Results first posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention): treatment as usual
- Self-monitoring for patients with Diabetes mellitus type 2 (Experimental): Patients are self-monitoring and submitting their vital parameters.
  Interventions: Other: Self-monitoring for patients with Diabetes mellitus type 2
- Nurse-monitoring for patients with Diabetes mellitus type 2 (Experimental): Nurses are measuring and entering the vital parameters of the patients.
  Interventions: Other: Nurse-monitoring for patients with Diabetes mellitus type 2

INTERVENTIONS:
Other: Self-monitoring for patients with Diabetes mellitus type 2 — Patients are submitting their vital parameters via a Web Portal or automatic devices to the hospital.
  Arms: Self-monitoring for patients with Diabetes mellitus type 2
Other: Nurse-monitoring for patients with Diabetes mellitus type 2 — Nurses are submitting the vital parameters of the patient via mobile device.
  Arms: Nurse-monitoring for patients with Diabetes mellitus type 2

SUMMARY:
Evaluation whether the introduction of large-scale personalized and technology supported telemonitoring and health coaching interventions produces benefits in terms of health related quality of life, health status and empowerment of patients with type 2 diabetes mellitus. In addition, the trials evaluate the economical and organizational impact of the new services and examine their acceptability by patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* T2DM diagnosed > 3 months prior to the enrollment
* HbA1c >= 6,5 %
* Capability of filling questionnaires by their own language
* Being able to use the devices provided
* Being cognitively able to participate

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Klinikum Klagenfurt, Klagenfurt, Carinthia
  - LKH Laas, Kötschach, Carinthia
  - LKH Villach, Villach, Carinthia

RESULTS

PARTICIPANT FLOW:
Groups:
- Nurse-monitoring for Patients With Diabetes Mellitus Type 2: nurse-monitoring for patients with Diabetes Mellitus
  Nurses are entering vital parameters of the patient with mobile devices
Period: Overall Study
Arm/Group | Control Group | Self-monitoring for Patients With Diabetes Mellitus Type 2 | Nurse-monitoring for Patients With Diabetes Mellitus Type 2
Started | 76 | 114 | 3
Completed | 61 | 101 | 0 (Due to high age and bad health conditions no patients finished (nursing))
Not Completed | 15 | 13 | 3

BASELINE CHARACTERISTICS:
Groups:
- Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2: Patients are self-monitoring and submitting their vital parameters.
  Self-monitoring for patients with Diabetes mellitus type 2: Patients are submitting their vital parameters via a Web Portal or automatic devices to the hospital.
  Nurses are measuring and entering the vital parameters of the patients.
  Nurse-monitoring for patients with Diabetes mellitus type 2: Nurses are submitting the vital parameters of the patient via mobile device.
  No patients using the mobile nursing finished the study, so in the final statistical analysis they were not analysed as separate arm.
  Due to low enrollement in the Nurse Monitoring arm, it is combined in this module.
- Total: Total of all reporting groups
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2 | Total
Number analyzed (Participants) | 76 | 117 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.38 (11.13) | 60.35 (11.68) | 61.54 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 55 | 86
  Male | 45 | 62 | 107
Region of Enrollment [Number; unit: participants]
  Austria | 76 | 117 | 193

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life as Measured by the Short Form 36 Version 2 Questionnaire
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status.
  Mearurement at the beginning and after 12 months, Scales from 0 to 100, higher values represent a better outcome; Data are mean scores (SD); differences between groups after 12 month were compared by using Mann-Whitney-U-tests.
Time Frame: 12 months
Population: No patients of the Nurse-Monitoring Group finished the study, as a consequence no SF36 after 12 months were delivered, so a calculation and evaluation for this group could not be conducted.
Measure: Mean (Standard Deviation); unit: units on a scale (General health score)
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 61 | 101
units on a scale (General health score)
  Physical Functioning 0-100 Score baseline | 69.2 (25.8) | 72.5 (25.2)
  Physical Functioning 0-100 Score | 74.9 (24.1) | 77.1 (22.3)
  Role Physical 0-100 Score baseline | 58.5 (29.5) | 63.8 (24.3)
  Role Physical 0-100 Score | 68.3 (29.3) | 72.5 (25.1)
  Bodily Pain 0-100 Score baseline | 59.8 (33.6) | 62.2 (31.0)
  Bodily Pain 0-100 Score | 66.7 (30.9) | 66.5 (30.0)
  General Health 0-100 Score baseline | 62.6 (19.3) | 62.2 (16.6)
  General Health 0-100 Score | 67.9 (17.9) | 69.4 (18.8)
  Vitality 0-100 Score baseline | 56.3 (25.7) | 58.4 (62.5)
  Vitality 0-100 Score | 61.6 (23.6) | 63.2 (19.1)
  Social Functioning 0-100 Score baseline | 80.1 (23.1) | 81.3 (22.1)
  Social Functioning 0-100 Score | 86.7 (18.8) | 81.3 (26.6)
  Role Emotional 0-100 Score baseline | 67.5 (28.2) | 70.7 (24.5)
  Role Emotional 0-100 Score | 77.7 (28.4) | 78.7 (25.3)
  Mental Health 0-100 Score baseline | 72.2 (21.7) | 72.1 (18.8)
  Mental Health 0-100 Score | 76.1 (19.6) | 72.6 (20.1)
  PCS Physical Component Score baseline | 43.7 (10.4) | 45.1 (9.9)
  PCS Physical Component Score | 46.3 (9.6) | 47.9 (9.5)
  MCS Mental Component Score baseline | 47.2 (11.9) | 47.9 (11.7)
  MCS Mental Component Score | 50.6 (11.9) | 49.1 (11.6)

2. Primary Outcome: HbA1c
Description: HbA1c was taken at the beginning of the study and after 12 months.
Time Frame: 12 months
Population: No patients of the Nurse-Monitoring Group finished the study, as a consequence no HbA1c after 12 months were delivered, so a calculation and evaluation for this group could not be conducted.
Measure: Mean (Standard Deviation); unit: HbA1c [%]
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 61 | 101
HbA1c [%]
  HbA1c values: first examination | 8.1 (1.2) | 8.7 (1.9)
  HbA1c values after 12 months | 7.5 (1.1) | 7.5 (1.5)
Statistical Analysis 1: Comparison: Control Group vs Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Blood Pressure
Time Frame: 12 months
Population: Not all Participants delivered data, reliable data was used. No patients of the Nurse-Monitoring Group finished the study, as a consequence no blood pressure after 12 months were delivered, so a calculation and evaluation for this group could not be conducted.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 54 | 77
mmHg
  diastolic baseline | 86.7 (12.9) | 88.9 (12.6)
  systolic baseline | 150.4 (21.3) | 153.7 (23.1)
  diastolic after 12 months | 85.2 (13.0) | 84.8 (12.6)
  systolic after 12 months | 149.3 (21.1) | 148.7 (23.6)
Statistical Analysis 1: Comparison: Control Group vs Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2; Blood pressure: diastolic; Test type: Superiority or Other; p = 0.182, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Blood Lipids
Time Frame: 12 months
Population: Not all Participants delivered reliable data; Measurements at the beginning of the trial and after 12 months; No patients of the Nurse-Monitoring Group finished the study, as a consequence no blood lipids after 12 months were delivered, so a calculation and evaluation for this group could not be conducted.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 56 | 81
mg/dL
  LDL Cholesterol after 12 months | 104.3 (38.7) | 107.6 (44.2)
  LDL Cholesterol baseline | 107.5 (36.3) | 112.1 (42.5)
  Cholesterol after 12 months | 185.2 (41.6) | 186.1 (51.3)
  Cholesterol after baseline | 186.8 (37.8) | 197.6 (53.1)
  HDL-cholesterol after 12 months | 51.3 (17.6) | 48.1 (16.9)
  HDL-cholesterol baseline | 48.2 (16.8) | 47.1 (12.6)

5. Secondary Outcome: Body Weight
Time Frame: 12 months
Population: baseline demographic characteristics; No patients of the Nurse-Monitoring Group finished the study, as a consequence no Body weight after 12 months were delivered, so a calculation and evaluation for this group could not be conducted.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 61 | 101
kilograms
  body weight baseline | 90.2 (19.0) | 90.74 (20.0)
  body weight after 12 months | 91.22 (19.32) | 91.64 (19.94)

6. Secondary Outcome: Medication Changes
Description: Insulin, Change? -> Yes/No
Time Frame: 12 months
Population: No data about medical changes could be analysed at the end of the study, no data were collected.
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Presence of Diabetic Complications
Time Frame: 12 months
Population: No data about the presence of diabetic complications could be analysed at the end of the study, no data was collected for this secondary outcome.
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Hospitalisations
Description: The number of inpatient stays comparing intervention and control group was conducted.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of inpatient stays
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Number analyzed (Participants) | 76 | 117
number of inpatient stays | 0.33 (0.63) | 0.38 (0.71)

ADVERSE EVENTS:
Groups:
- Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2: Patients are self-monitoring and submitting their vital parameters.
  Self-monitoring for patients with Diabetes mellitus type 2: Patients are submitting their vital parameters via a Web Portal or automatic devices to the hospital.
  Home nursing is also included. Nurses are measuring and entering the vital parameters of the patients.
  Nurse-monitoring for patients with Diabetes mellitus type 2: Nurses are submitting the vital parameters of the patient via mobile device.
  No patients using the mobile nursing finished the study, so in the final statistical analysis they were not analysed as separate arm.
  Due to low enrollement in the Nurse Monitoring arm, it is combined in this module.
Arm/Group | Control Group | Self-monitoring and Nurse Monitoring Diabetes Mellitus Type 2
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/101
Other Adverse Events (participants affected / at risk) | 0/61 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes